CLINICAL TRIAL: NCT03099577
Title: Phase I Study of PET/CT-directed Hyperfractionated Radiation Dose Escalation With Concurrent Weekly Carboplatin and Paclitaxel in Stage III Non-small Cell Lung Cancer
Brief Title: PET/CT-directed Hyperfractionated Radiation Dose Escalation in Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, director,department of radiation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGH201708
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- radiochemotherapy 1 (Experimental): Patients will be treated with radiation therapy 64.8 Gy
  Interventions: Radiation: radiochemotherapy 1
- radiochemotherapy 2 (Experimental): Patients will be treated with radiation therapy 69.6 Gy
  Interventions: Radiation: radiochemotherapy 2
- radiochemotherapy 3 (Experimental): Patients will be treated with radiation therapy 74.4 Gy
  Interventions: Radiation: radiochemotherapy 3
- radiochemotherapy 4 (Experimental): Patients will be treated with radiation therapy 79.2 Gy
  Interventions: Radiation: radiochemotherapy 4
- radiochemotherapy 5 (Experimental): Patients will be treated with radiation therapy 84 Gy
  Interventions: Radiation: radiochemotherapy 5
- radiochemotherapy 6 (Experimental): Patients will be treated with radiation therapy 88.8 Gy
  Interventions: Radiation: radiochemotherapy 6
- radiochemotherapy 7 (Experimental): Patients will be treated with radiation therapy 93.6 Gy
  Interventions: Radiation: radiochemotherapy 7

INTERVENTIONS:
Radiation: radiochemotherapy 1 — concurrent radiochemotherapy: radiotherapy dose level 1: 60 Gy at 2 Gy/Fx/d, then 4.8 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 1
  Arms: radiochemotherapy 1
Radiation: radiochemotherapy 2 — concurrent radiochemotherapy: radiotherapy dose level 2: 60 Gy at 2 Gy/Fx/d, then 9.6 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 2
  Arms: radiochemotherapy 2
Radiation: radiochemotherapy 3 — concurrent radiochemotherapy: radiotherapy dose level 3: 60 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 3
  Arms: radiochemotherapy 3
Radiation: radiochemotherapy 4 — concurrent radiochemotherapy: radiotherapy dose level 4: 60 Gy at 2 Gy/Fx/d, then 19.2 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 4
  Arms: radiochemotherapy 4
Radiation: radiochemotherapy 5 — concurrent radiochemotherapy: radiotherapy dose level 5: 60 Gy at 2 Gy/Fx/d, then 4.8x5 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 5
  Arms: radiochemotherapy 5
Radiation: radiochemotherapy 6 — concurrent radiochemotherapy: radiotherapy dose level 6: 60 Gy at 2 Gy/Fx/d, then 4.8x6 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 6
  Arms: radiochemotherapy 6
Radiation: radiochemotherapy 7 — concurrent radiochemotherapy: radiotherapy dose level 7: 60 Gy at 2 Gy/Fx/d, then 4.8x7 Gy at 1.2 Gy/Fx/bid concurrent concurrent chemotherapy :carboplatin area under the curve (AUC) 2; paclitaxel: 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen 7
  Arms: radiochemotherapy 7

SUMMARY:
The goal of this study is to find the maximum tolerable dose of radiation that can be delivered combined with chemotherapy (carboplatin & paclitaxel) in patients with stage III non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard of care for unresectable stage III NSCLC based on the results of phase III randomised trials. The current standard radiation therapy dose has remained 60- Gy at -2 Gy/fraction for nearly four decades (60Gy), with local disease control rates of approximately 50% and a median overall survival of only 18 months.These results are suboptimal and more effective treatment regimens are needed.

We hypothesize that hyperfractionated radiation dose escalation to residual tumor volumes after standard chemoradiotherapy as defined by positron emission tomography (PET) /computed tomography (CT) would improve local control and overall survival while reducing the acute and late normal tissue toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have FDG-avid and histologically or cytologically proven non-small cell lung cancer.
2. Age 1 8-75.
3. Zubrod performance status 0-2.
4. Stage III ( American Joint Committee on Cancer AJCC, 7th ed.).
5. No prior radiation to the thorax that would overlap with the current treatment field.
6. Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </=1 .5 times ULN.
7. A signed informed consent must be obtained prior to therapy.
8. Induction chemotherapy is allowed.
9. Life expectancy more than 3 months.

Exclusion Criteria:

1. Patients with any component of small cell lung carcinoma are excluded from this study.
2. Patients with evidence of a malignant pleural or pericardial effusion are excluded.
3. Prior radiotherapy that would overlap the radiation fields.
4. Uncontrolled concurrent illness including, but not limited to: Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.
5. Known hypersensitivity to paclitaxel.
6. Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
7. Acquired Immune Deficiency Syndrome.
8. Conditions precluding medical follow-up and protocol compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
  Maximum Tolerated Dose is defined as CTCAE 4 grade 3 acute radiation-related toxicity

SECONDARY OUTCOMES:
Time to Local Failure | 2 years
  Local control will be assessed radiographically using endoscopy with biopsy and a positron emission computed tomography-CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Principal Investigator — the ethic committee of shanghai genernal hospital
Locations (1):
- the Ethic Committee of Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No